CLINICAL TRIAL: NCT02904538
Title: Perineural Versus Systemic Dexamethasone to Prolong Regional Anesthesia in Front Foot Surgery
Acronym: ADRIATIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0277; 2016-001341-41 (Other: 2016-001341-41)
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Pain Management After Surgery
Keywords: Dexamethasone; Regional anesthesia; Front foot surgery; Metacarpal osteotomy
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Perineural group (Experimental): 1cc (4mg) of dexamethasone will be administrated in perineural injection. 2.5cc of isotonic saline solution will be administrated in systemic injection.
  Interventions: Drug: Dexamethasone
- systemic group (Experimental): 1cc of isotonic saline will be administrated in perineural injection. 2.5cc (10mg) of dexamethasone will be administrated in systemic injection.
  Interventions: Drug: Dexamethasone; Drug: isotonic saline

INTERVENTIONS:
Drug: Dexamethasone
Drug: isotonic saline
  Arms: systemic group

SUMMARY:
Both perineural and systemic dexamethasone administration allows an increase in analgesic duration of regional anesthesia.

There is a lack of data to determine wich route allows a longer analgesic effect.

This study aims to determine wether perineural dexamethasone allows a longer analgesic duration than systemic route in combination with regional anesthesia (Ropivacaine 0.375%) for front foot surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind controlled trial.

All Patients undergoing front foot surgery with metacarpal osteotomy will be screened for inclusion in the protocol. All patients without exclusion criteria will be included in the study.

All patients will receive 30cc mixure of Ropivacaine 0,375% in perineural injection and surgery will be performed under regional anesthesia only. If needed, a sedation with midazolam (1mg) will be performed.

The patients will be randomized over 2 groups:

* "Perineural group":

  * 1cc (4mg) of dexamethasone will be administrated in perineural injection
  * 2.5cc of isotonic saline solution will be administrated in systemic injection
* "Systemic group":

  * 1cc of isotonic saline will be administrated in perineural injection
  * 2.5cc (10mg) of dexamethasone will be administrated in systemic injection

For both groups perineural injection will be performed at the ankle and the following nerves will be targeted: the tibial nerve, saphenous nerve, the deep fibular nerve, the superficial fibular nerve and the sural nerve.

Post-operative analgesia will be reached with paracetamol (1gr each 6 hours) and Ketoprofen (100mg each 12 hours).

After surgery, patients will be asked to write down the time to the first opioids request during the first 48 hours, maximal pain during the first 48H using a visual analog scale, occurrence of nausea or vomiting, overall satisfaction regarding pain relief management and any significant side effects during the first 7 days.

The primary objective of the study is to determine if perineural dexamethasone is associated with a longer analgesic duration than systemic route in combination with regional anesthesia (Ropivacaine 0.375%) for front foot surgery.

The primary end-point will be time to the first opioids request during the first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* front foot surgery with metacarpal osteotomy under regional anesthesia
* >18 years old
* consent to participate in the study

Exclusion Criteria:

* refusal to participate
* pregnancy
* feeding
* pre existing neuropathy
* ropivacaine allergy
* paracetamol allergy
* liver failure
* cardiac failure
* ketoprofen allergy
* gastric ulcer within the previous year
* tramadol allergy
* history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
time to the first opioids request | during the first 48 hours

SECONDARY OUTCOMES:
occurrence of nausea or vomiting | at day 1
  during the first 48 hours
overall satisfaction regarding pain relief management | at day 1
  overall satisfaction regarding pain relief management (using following questionnaire : No pain - Light pain - Moderate pain - Significant pain - Excruciating pain)
any significant side effects | during the first 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Marty P, Rontes O, Chassery C, Vuillaume C, Basset B, Merouani M, Marquis C, Bataille B, Chaubard M, Mailles MC, Ferre F, Delbos A. Perineural Versus Systemic Dexamethasone in Front-Foot Surgery Under Ankle Block: A Randomized Double-Blind Study. Reg Anesth Pain Med. 2018 Oct;43(7):732-737. doi: 10.1097/AAP.0000000000000769. PMID 29630032